CLINICAL TRIAL: NCT05616975
Title: Reliability, Validity, Normative Data, and Accuracy of SWAY Mobile Application Assessments in Healthy Adults
Brief Title: SWAY Mobile Application Assessments in Healthy Adults
Status: Withdrawn | Type: Observational
Why Stopped: This project never entered the recruitment phase due to issues with hiring study personnel.
Sponsor: University of Oklahoma (Other)
Collaborators: SWAY Medical, Inc (Unknown); College of Medicine Alumni Association (Unknown); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Sponsor
Other Study IDs: OU IRB 14031
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Reliability; Validity; Normative Data
Keywords: reliability; validity; normative data; balance assessments; functional assessments; cognitive assessments
MeSH Terms: interventions — Reproducibility of Results

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- reliability: Assessing the test-retest reliability of SWAY Balance, Functional, and Cognitive tests
  Interventions: Other: test-retest reliability
- validity: Investigating the construct validity of SWAY Balance, Functional, and Cognitive tests
  Interventions: Other: construct validity
- normative: Collection of normative SWAY Balance, Functional, and Cognitive data
  Interventions: Other: normative data

INTERVENTIONS:
Other: test-retest reliability — Assessing the test-retest reliability of SWAY Balance, Functional, and Cognitive tests.
  Groups: reliability
Other: construct validity — Investigating the construct validity of SWAY Balance, Functional, and Cognitive tests.
  Groups: validity
Other: normative data — Collection of normative SWAY Balance, Functional, and Cognitive data.
  Groups: normative

SUMMARY:
SWAY Medical, Inc. (SWAY) has developed a mobile application that assesses balance, functional performance, and cognitive function. Clinical reliability, validity, and normative data have been studied extensively in individuals aged 5 to 20. The accuracy of the SWAY Mobile Application in assessing conditions associated with head injury has also been well established. The objectives of this study are to examine the reliability and validity, and establish normative data, for SWAY balance, functional, and cognitive assessments in healthy adults aged 21-90. The SWAY smartphone app will be used to record balance, simple reaction time, impulse control, inspection time, working memory, reverse number counting, flanker task, modified Stroop, and 30 second chair stand test results. The following tests will be administered to participants: Test of Premorbid Functioning, WAIS-IV Logical Memory, WMS-IV Older Adult Logical Memory, Animal Fluency, Boston Naming Test, D-KEFS Color Word Interference Test, WMS-IV Symbol Span, WAIS-IV Coding, Auditory Consonant Trigrams, Verbal Fluency (FAS), and Flanker Inhibitory Control and Attention Test.

DETAILED DESCRIPTION:
Specific Aims The objectives of this study are to examine the reliability and validity, and to establish normative data, for SWAY balance, functional, and cognitive assessments in healthy adults aged 21-90.

Aim 1, Hypothesis 1: Sway balance, functional, and cognitive test scores collected at baseline and 30 days will show acceptable test-retest reliabilities.

Aim 2, Hypothesis 2: Sway balance, functional, and cognitive test scores will have medium correlations with psychometrically supported neuropsychological tests of similar constructs (convergent validity) and small correlations with psychometrically supported neuropsychological tests of disparate constructs (discriminant validity).

Aim 3, Hypothesis 3: Sway balance, functional, and cognitive normative test scores will vary significantly across age, education, sex, and race.

ELIGIBILITY:
Exclusion Criteria:

* Uncorrected visual or hearing impairment that interferes with testing
* Alcohol or drug intoxication
* Severe, untreated psychiatric illness (e.g., schizophrenia, bipolar disorder, depression)
* Cognitive impairment (e.g. dementia)
* Motor impairments that may interfere with testing
* Individuals who have a self-reported history of falling or are believed to be at-risk of falling may be excluded from the balance testing portion of the study but will remain eligible to participate in the functional and cognitive assessment portions of the study. Participants over the age of 50 will complete a short fall risk screening assessment.
* Individuals who have a musculoskeletal injury affecting functional movement and balance may be excluded from the balance testing portion of the study but will remain eligible to participate in the cognitive assessment portions of the study.
* Volunteers may also be excluded from portions of this study if they do not have the necessary technology to maintain a Zoom connection required for remotely administered follow-up assessments, and a smart-device capable of downloading and operating the SWAY application.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants:
  Not less than seven hundred (700) and up to one thousand (1000) men and women from the University of Oklahoma. OU students, residents, staff, faculty, and patients will be recruited through flyers posted and distributed on campus, in clinics, on social media and through emails. Additional participants will be recruited from the community as needed via flyers distributed at local hospitals, clinics, senior living facilities, and through newspaper and radio advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Balance Assessments | <15 minutes
  i. Modified balance error scoring system protocol (mBESS) in individuals less than 55 years of age ii. CDC 4-stage Balance test for individuals greater than or equal to 55 years of age
Functional Assessments | <15 minutes
  i. SWAY 30 Second Chair Stand Test (functional)
Cognitive Assessments | 15 minutes
  i. SWAY Memory (visual working memory) ii. SWAY Modified Erikson Flanker Task (visual scanning) iii. SWAY Simple Reaction Time (visual simple RT) iv. SWAY Impulse Control (visual go/no-go) v. SWAY Inspection Time (visual processing speed/reaction time) vi. SWAY Number Counting (visual processing speed) vii. SWAY Modified Stroop Test (executive function)